CLINICAL TRIAL: NCT01020357
Title: Long-Term Effects On Sleep Of Methylxanthine Therapy For Apnea Of Prematurity
Brief Title: Caffeine for Apnea of Prematurity-Sleep (CAP-S) Study
Acronym: CAP-S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIH-R01HL098045; R01HL098045 (NIH)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Apnea of Prematurity
Keywords: preterm infants; very low birthweight; apnea of prematurity; methylxanthines; sleep disturbance; obstructive sleep apnea syndrome; polysomnography; sleep disruption
MeSH Terms: conditions — Apnea; Parasomnias; Sleep Apnea, Obstructive | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- caffeine (Active Comparator)
  Interventions: Drug: Caffeine citrate injection
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Caffeine citrate injection — Loading dose: 20 mg/kg administered over at least 30 minutes via IV infusion or over at least 10 minutes via slow IV injection.
  Daily maintenance dose (to commence at least 24 hours after loading dose): 5 mg/kg, administered over at least 10 minutes via IV infusion, or over at least 5 minutes via slow IV injection. Maintenance dose to be adjusted for body weight every 7 days. If indicated, maintenance dose may be increased to a maximum of 10 mg/kg. May be given orally once full enteral feeds are established.
  Duration of treatment: discontinue after infant has tolerated at least 5 consecutive days without positive pressure support AND when the infant is judged by the attending clinician to be no longer a candidate for methylxanthine therapy.
  Other Names: CafCit
  Arms: caffeine
Drug: placebo — normal saline
  Arms: placebo

SUMMARY:
Apnea of prematurity is a common condition that is usually treated with methylxanthines. Methylxanthines are adenosine receptor blockers that have powerful influences on the central nervous system. However, little is known about the long-term effects of methylxanthines on the developing brain.

The Caffeine for Apnea of Prematurity-Sleep (CAP-S) Study is a sub-study of the main Caffeine for Apnea of Prematurity (CAP) trial, an international placebo-controlled randomized trial of methylxanthine therapy for apnea of prematurity. This sub-study is designed to take advantage of this cohort of ex-premature, 5-7 year old children who were randomized at birth to receive either caffeine or placebo, and are currently receiving detailed neurocognitive and behavioral assessments in the CAP trial.

DETAILED DESCRIPTION:
The use of methylxanthines as therapy for apnea of prematurity may be a double-edged sword. Although widely-used, and efficacious for treatment of apnea of prematurity, long-term drug effects have not been rigorously studied. Neonatal methylxanthine therapy may have long-term impacts on sleep organization and ventilatory control. The CAP trial, funded by the Canadian Institutes of Health Research, was initiated due to the paucity of well-controlled data on the long-term effects of methylxanthines in preterm infants. The initial CAP trial was a multicenter, randomized, placebo-controlled trial of caffeine vs placebo as treatment for apnea of prematurity with follow-up to a corrected age of 18 months. 2,006 infants were enrolled. The CAP trial found that methylxanthines reduced the rates of bronchopulmonary dysplasia (BPD) and cerebral palsy (CP), and did not affect mortality. However, concerns remain regarding long-term sequelae of methylxanthine use. The Canadian Institutes of Health Research have therefore funded further follow-up of the entire CAP trial cohort to age 5 years, corrected for prematurity. The key objectives of this study are to examine the impact of methylxanthines on neurocognition and behavior. This ongoing parent study provides an opportunity to determine potential long-term effects of methylxanthines on sleep disorders, and to correlate these findings with daytime functioning. Our overall hypothesis is that methylxanthine use in preterm infants, while beneficial in the short term, results in longstanding abnormalities in the regulation of sleep, and breathing during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 5-7 years who are enrolled in the CAP trial.
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Aim 1: The primary outcome is the mean actual sleep time as measured by actigraphy, between subjects who received caffeine vs placebo. | 5-7 years
Aim 2: The primary outcome is the apnea hypopnea index (AHI) between subjects who received caffeine vs placebo. | 5-7 years
Aim 3: The primary outcome is the correlation between full-scale IQ from the Wechsler Preschool and Primary Scale of Intelligence (measured in the CAP trial rather than directly from this protocol), sleep time and AHI. | 5-7 years

SECONDARY OUTCOMES:
Questionnaire data: National Sleep Foundation (NSF) and Pediatric Sleep Questionnaire (PSQ) scores | 5-7 years
Polysomnography data: Sleep architecture, arousal index, central apnea index, SpO2 and periodic limb movement index. | 5-7 years

CONTACTS AND LOCATIONS:
Overall Officials: Carole Marcus, M.B.B.Ch., Principal Investigator — University of Pennsylvania
Locations (4):
- Australia (2):
  - Mercy Hospital for Women, Melbourne
  - Royal Women's Hospital, Melbourne
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Result] Marcus CL, Meltzer LJ, Roberts RS, Traylor J, Dix J, D'ilario J, Asztalos E, Opie G, Doyle LW, Biggs SN, Nixon GM, Narang I, Bhattacharjee R, Davey M, Horne RS, Cheshire M, Gibbons J, Costantini L, Bradford R, Schmidt B; Caffeine for Apnea of Prematurity-Sleep Study. Long-term effects of caffeine therapy for apnea of prematurity on sleep at school age. Am J Respir Crit Care Med. 2014 Oct 1;190(7):791-9. doi: 10.1164/rccm.201406-1092OC. PMID 25171195
- [Result] Marcus CL, Traylor J, Biggs SN, Roberts RS, Nixon GM, Narang I, Bhattacharjee R, Davey MJ, Horne RS, Cheshire M, Gibbons KJ, Dix J, Asztalos E, Doyle LW, Opie GF, D'ilario J, Costantini L, Bradford R, Schmidt B. Feasibility of comprehensive, unattended ambulatory polysomnography in school-aged children. J Clin Sleep Med. 2014 Aug 15;10(8):913-8. doi: 10.5664/jcsm.3970. PMID 25126039